CLINICAL TRIAL: NCT04998201
Title: A Double-Blind, Placebo-Controlled Phase 2b Study to Evaluate the Efficacy and Safety of ARO-APOC3 in Adults With Mixed Dyslipidemia
Brief Title: Study of ARO-APOC3 in Adults With Mixed Dyslipidemia
Acronym: MUIR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AROAPOC3-2002; 2021-000688-57 (EudraCT Number)
Record Dates: First submitted 2021-08-03; First posted 2021-08-10 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Mixed Dyslipidemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- ARO-APOC3 10 mg, Day 1 and Week 12 (Experimental): 2 doses of ARO-APOC3 by subcutaneous (sc) injection
  Interventions: Drug: ARO-APOC3
- ARO-APOC3 25 mg, Day 1 and Week 12 (Experimental): 2 doses of ARO-APOC3 by subcutaneous (sc) injection
  Interventions: Drug: ARO-APOC3
- ARO-APOC3 50 mg, Day 1 and Week 12 (Experimental): 2 doses of ARO-APOC3 by subcutaneous (sc) injection
  Interventions: Drug: ARO-APOC3
- ARO-APOC3 50 mg, Day 1 and Week 24 (Experimental): 2 doses of ARO-APOC3 by subcutaneous (sc) injection
  Interventions: Drug: ARO-APOC3
- Placebo, Day 1 and Week 12 or Week 24 (Placebo Comparator): calculated volume to match active treatment by sc injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ARO-APOC3 — ARO-APOC3 Injection
  Arms: ARO-APOC3 10 mg, Day 1 and Week 12; ARO-APOC3 25 mg, Day 1 and Week 12; ARO-APOC3 50 mg, Day 1 and Week 12; ARO-APOC3 50 mg, Day 1 and Week 24
Drug: Placebo — Sterile Normal Saline (0.9% NaCl)
  Arms: Placebo, Day 1 and Week 12 or Week 24

SUMMARY:
Participants who have met all protocol eligibility criteria will be randomly assigned to treatment (ARO-APOC3 or placebo) in a double-blind fashion and will be evaluted for safety and efficacy over 48 weeks. Participants will be counseled to remain on a specified diet throughout the study, as recommended by the Investigator in accordance with local standard of care. After week 48, participants will be eligible and invited to consent and continue in an open-label extension study. All placebo participants who opt to continue will switch to active drug (ARO-APOC3) during the extension study.

ELIGIBILITY:
Inclusion Criteria:

Based on medical history, evidence of TG ≥ 150 mg/dL but ≤ 499 mg/dL on more than one occasion

* Fasting levels at Screening of non-HDL-C ≥ 100 mg/dL OR LDL-C ≥ 70 mg/dL after at least 4 weeks of stable diet and stable optimal statin therapy
* Mean fasting TG ≥ 150 mg/dL and ≤ 499 mg/dL during Screening collected at two separate and consecutive visits and at least 7 days apart and not more than 14 days apart
* Willing to follow diet counseling as per Investigator judgment based on local standard of care
* Participants of childbearing potential (males & females) must use highly-effective contraception during the study and for at least 24 weeks following the last dose of study medication. Males must not donate sperm and females must ot donate eggs during the study and for at least 24 weeks following the last dose of study medication.
* Women of childbearing potential must have a negative pregnancy test at Screening and cannot be breastfeeding
* Women of childbearing potential on hormonal contraceptives must be stable on the medication for ≥ 2 menstrual cycles prior to Day 1
* Willing to provide written informed consent and to comply with study requirements

Exclusion Criteria:

* Current use or use within 365 days from Day 1 of any hepatocyte targeted siRNA or antisense oligonucleotide molecule
* Active pancreatitis within 12 weeks prior to Day 1
* Any planned bariatric surgery or similar procedures to induce weight loss from consent through end of study
* Acute coronary syndrome event within 24 weeks of Day 1
* Major surgery within 12 weeks of Day 1
* Planned coronary intervention (e.g., stent placement or heart bypass) during the study
* New York Heart Association Class II, III or IV heart failure or last known ejection fraction of <30%
* Uncontrolled hypertension
* Known history of human immunodeficiency virus (HIV) infection, seropositive for Hepatitis B (HBV), seropositive for Hepatitis C (HCV)
* Uncontrolled hypothyroidism or hyperthyroidism
* Hemorrhagic stroke within 24 weeks of Day 1
* History of bleeding diathesis or coagulopathy
* Current diagnosis of nephrotic syndrome
* Systemic use of corticosteroids or anabolic steroids within 4 weeks prior to Day 1 or planned use during the study
* Malignancy within the last 2 years prior to date of consent requiring systemic treatment (some exceptions apply)

Note: additional inclusion/exclusion criteria may apply per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
Percent Change from Baseline in Fasting Triglycerides (TG) at Week 24 | Baseline, Week 24

SECONDARY OUTCOMES:
Percent Change from Baseline in Fasting TG | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 36, Week 48
Percent Change from Baseline in Apolipoprotein (APO) C-III at Week 24 | Baseline, Week 24
Percent Change from Baseline in APOC-III Over Time | Baseline, up to Week 48
Percent Change from Baseline in Fasting Non High Density Lipoprotein Cholesterol (Non-HDL-C) at Week 24 | Baseline, Week 24
Percent Change form Baseline in Non-HDL-C Over Time | Baseline, up to Week 48
Percent Change from Baseline in Fasting High Density Lipoprotein Cholesterol (HDL-C) at Week 24 | Baseline, Week 24
Percent Change from Baseline in HDL-C Over Time | Baseline, up to Week 48
Percent Change from Baseline in Fasting Total Apolipoprotein B (ApoB) at Week 24 | Baseline, Week 24
Percent Change from Baseline in ApoB Over Time | Baseline, up to Week 48
Percent Change from Baseline in Fasting Total Low Density Lipoprotein Cholesterol (LDL-C) Using Ultracentrifugation at Week 24 | Baseline, Week 24
Percent Change from Baseline in Fasting Total LDL-C Using Ultracentrifugation Over Time | Baseline, up to Week 48
Number of Participants with Treatment-Emergent Adverse Events (AEs) and/or Serious Adverse Events (SAEs) at Week 24 | Week 24
Number of Participants with Treatment- Emergent AEs and/or SAEs Through Week 48 | up to Week 48
Change from Baseline in Plasma Concentrations of ARO-APOC3 Over Time | up to Week 24
Pharmacokinetics (PK) of ARO-APOC3: Maximum Observed Plasma Concentration (Cmax) | up to Week 24
PK of ARO-APOC3: Time to Maximum Plasma Concentration (Tmax) | up to Week 24
PK of ARO-APOC3: Area Under the Plasma Concentration Versus Time Curve From Zero to Time of Last Measurable Concentration (AUClast) | up to Week 24

CONTACTS AND LOCATIONS:
Locations (30):
- United States (15):
  - Research Site 3, Beverly Hills, California
  - Research Site 8, Northridge, California
  - Research Site 2, Boca Raton, Florida
  - Research Site 1, Fort Lauderdale, Florida
  - Research Site 14, Miami Springs, Florida
  - Research Site 5, Pembroke Pines, Florida
  - Research Site 18, Dunwoody, Georgia
  - Research Site 31, Las Vegas, Nevada
  - Research Site 17, New Windsor, New York
  - Research Site 12, Dayton, Ohio
  - Research Site 4, Franklin, Ohio
  - Research Site 7, Greenville, South Carolina
  - Research Site 6, Houston, Texas
  - Research Site 32, Houston, Texas
  - Research Site 13, San Antonio, Texas
- Australia (4):
  - Research Site 30, Morayfield, Queensland
  - Research Site 29, Adelaide, South Australia
  - Research Site 19, Clayton, Victoria
  - Research Site 27, Joondalup, Western Australia
- Canada (2):
  - Research Site 15, Concord, Ontario
  - Research Site 10, Montreal, Quebec
- Hungary (3):
  - Research Site 20, Balatonfüred
  - Research Site 21, Debrecen
  - Research Site 22, Nyíregyháza
- New Zealand (2):
  - Research Site 11, Auckland
  - Research Site 16, Christchurch
- Poland (4):
  - Research Site 28, Lodz
  - Research Site 24, Lodz
  - Research Site 25, Poznan
  - Research Site 26, Rzeszów

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ballantyne CM, Vasas S, Azizad M, Clifton P, Rosenson RS, Chang T, Melquist S, Zhou R, Mushin M, Leeper NJ, Hellawell J, Gaudet D. Plozasiran, an RNA Interference Agent Targeting APOC3, for Mixed Hyperlipidemia. N Engl J Med. 2024 Sep 12;391(10):899-912. doi: 10.1056/NEJMoa2404143. Epub 2024 May 28. PMID 38804517